CLINICAL TRIAL: NCT03125850
Title: Comparative Study of Psychology and Glaucoma Knowledge in Glaucoma Day-ward Patients Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mingkai Lin, chief physician, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Zhongshan OC
Record Dates: First submitted 2017-04-16; First posted 2017-04-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Glaucoma
Keywords: knowledge; psychology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- day-ward group (Experimental)
  Interventions: Other: randomized to day ward
- inpatient group (Active Comparator)
  Interventions: Other: randomized to inpaitent

INTERVENTIONS:
Other: randomized to day ward — Participants will be randomized to day-ward group, and will accept routine treatment, care, centralized education of glaucoma knowledge
  Arms: day-ward group
Other: randomized to inpaitent — Participants will be randomized to day-ward group, and will accept routine treatment, care, centralized education of glaucoma knowledge
  Arms: inpatient group

SUMMARY:
This study will compare the glaucoma day-ward patients' efficacy with inpatients by evaluating the glaucoma knowledge and psychology , and will analysis the reasons of the differences. Half of participants will receive treatment in day-ward, while the other half will receive treatment in hospital.

DETAILED DESCRIPTION:
Ophthalmic surgery has short operative time, quick recovery, and small anesthesia risk, making day case surgery the main management mode of ophthalmic surgery. This study will explore the differences of psychology and glaucoma knowledge between glaucoma day-ward patients and the inpatients. The data will be collected by scale on admission and discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with glaucoma;
2. Will receive glaucoma surgery;
3. Voluntary participation in this study;
4. Have enough language comprehension ability;
5. Best corrected visual acuity reach 0.1 or better;
6. Patient or his legal representative has sign the informed consent.

Exclusion Criteria:

1. Patient with mental disorder;
2. There are important viscera function failure or other serious disease, including clinical related coronary artery disease, cardiovascular disease or myocardial infarction into the group of the first six months; serious neurological or psychiatric illness; serious infections; coagulant function abnormality; general active infectious diseases; malignant tumor; serious immune diseases;
3. Patient with monocular blindness;
4. Axial length≤20 mm;
5. With other serious eye diseases;
6. Neurologic diseases that could affect the visual field;
7. 3 months prior to research to participate in any clinical study;
8. Researchers think not suitable to participate in this clinical trial subjects;
9. Refused to sign the informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Change of depression and anxiety score | at baseline and 1 hour before discharge
  The outcome will be measured by The Hospital Depression and Anxiety Scale (HADS). It consists of two subscales: HDAS-anxiety and HADS-depression. Each item is srored from 0-3, with higher scores indicating a higher level of depression and anxiety. For each of the seven-item subscales, the minimum sum score is 0, and the maximum is 21.
Change of glaucoma knowledge score | at baseline and 1 hour before discharge
  The outcome will be measured by The Gray Glaucoma Knowledge Questionaire. This quesionanire has a total maximum score of 17, with higher scores representing better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Lin, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-San University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-San Univerdity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No.